CLINICAL TRIAL: NCT05880667
Title: Adaptive Radiation for Abdominopelvic Metastases (ARAM)
Brief Title: Adaptive Radiation for Abdominopelvic Metastases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT-218; 23-1012 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Neoplasm - Soft Tissue Pelvis Malignant Secondary; Malignant Neoplasm of Stomach
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adaptive Stereotactic Body Radiation (Experimental): Simulation and treatment to be performed over 3-4 weeks per dose escalation
  Interventions: Radiation: Adaptive Stereotactic Body Radiation

INTERVENTIONS:
Radiation: Adaptive Stereotactic Body Radiation — Radiation therapy is given following generation of planning imaging at the time of simulation. A recent development has been diagnostic quality onboard imaging incorporated within radiation treatment machines. The incorporation of onboard imaging into standard practice has allowed the use Stereotactic Body Radiation (SBRT), which is a precise radiation technique that allows safe delivery of ablative radiation doses.
  More recently, the development of improved technologies and software have allowed radiation plans to be generated and delivered that are specific to the anatomy of the very moment the patient is being treated. This novel ability to adjust the radiation treatment plan based upon real time imaging is termed adaptive radiation therapy. This study will utilize the novel adaptive radiation therapy technology in a patient population with technically challenging disease to deliver ablative radiation with an appropriately low toxicity rate.

SUMMARY:
Single arm Phase I trial of adaptive stereotactic body radiation (SBRT) for abdominopelvic metastases. Adaptive SBRT will allow for escalation of the prescription dose and target coverage while maintaining grade 3+ toxicity no greater than 10%. Subjects with metastatic cancer to the abdomen or pelvis requiring local control or palliation will be enrolled.

DETAILED DESCRIPTION:
This is a dose-escalation study where the objective is to find the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of adaptive SBRT for abdominopelvic SBRT. There are 3 doses of interest 8Gy/fraction (level 1), 9Gy/fraction (level 2), and 10Gy/fraction (level 3). The starting dose will be level 2. We will use a Bayesian Optimal Interval Design (BOIN) to define dose escalation and de-escalation rules based on the proportion of patients experiencing a dose-limiting toxicity (DLT). DLT events are Grade 3 events possibly, probably, or definitely related to the study intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically or cytologically confirmed cancer that is metastatic (all solid tumor types accepted), with at least one target lesion untreated by radiation, IR techniques, or growing in the abdomen or pelvis. Adjacent lymph nodes in the same region (5 cm or closer) constitute one active lesion. Target lesion must be measurable according to RECIST v 1.1. Previous systemic therapies are allowed.
2. Age > 18 years.
3. ECOG performance status 0 or 1
4. Estimated survival of >/= 12 months
5. Subjects must have normal organ and marrow function as defined below

   * Absolute neutrophil count > 1,500/mcL
   * Platelets > 100,000/mcL
   * Total bilirubin < 2 mg/dL
   * AST/ALT (SGOT/SGPT) < 5X ULN
   * Creatinine < 1.5X ULN OR
   * Creatinine clearance ≥ 50 ml/min/1.73 m2 for subjects with creatinine levels above institutional normal
6. Subjects must possess the ability to understand and willingness to sign a written informed consent and HIPAA consent document. Translation services including translation of informed consent documents will be provided, as feasible, to encourage diversity of inclusion of eligible patients.

Exclusion Criteria:

1. Subjects must not be experiencing toxicity due to prior therapy that has not resolved to ≤Grade 1 by study registration, with the exception of sensory neuropathy related to previous systemic therapy exposure, alopecia and fatigue.
2. Subjects must not be receiving any other investigational agents.
3. Subjects must not have known peritoneal carcinomatosis visible on imaging.
4. Subjects must not have known active solid tumors on imaging outside of abdomen/pelvis noted on screening imaging
5. Subjects must not have 6 or more active metastatic sites.
6. Subjects must not have had prior radiotherapy to any target metastatic lesion. Prior radiotherapy to non-target sites is allowed.
7. Subjects must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Any condition or significant co-morbidity that prevents safe delivery of SBRT per the discretion of the treating physician(s).
9. Subjects must not be pregnant or breast-feeding. Refer to section 4.4 for further detail.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
To assess the ability of adaptive SBRT to deliver increased doses of radiation safely to patients with challenging anatomical locations of metastatic disease without causing unacceptable toxicity. | 3 months
  Cohorts of size 10 will be enrolled, Severe (grade 3) toxicity occurring within 3 months of treatment that is possibly, probably, or definitely related to trial therapy will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Meyer, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No